CLINICAL TRIAL: NCT04156867
Title: Evaluation of Outcomes of Discectomy With Dynesys in Treatment of Lumbar Disc Herniation: a Prospective Study
Brief Title: Evaluation of Outcomes of Discectomy With Dynesys in Treatment of Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY201410933-56
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Orthopedic Disorder of Spine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- simple discectomy (Experimental): traditional simple discectomy
  Interventions: Device: Dynesys

INTERVENTIONS:
Device: Dynesys — discectomy with Dynesys

SUMMARY:
To explore the clinical outcomes of discectomy with dynamic neutralization system(Dynesys) on treatment of single-segmental lumbar disc herniation(LDH) versus simple discectomy.

DETAILED DESCRIPTION:
The study was to explore the clinical outcomes of discectomy with dynamic neutralization system(Dynesys) on treatment of single-segmental lumbar disc herniation(LDH) versus simple discectomy. 128 patients with single-segmental LDH were randomly divided into discectomy with Dynesys group(group A) and simple discectomy group(group B). Both groups were evaluated by Visual Analogue Score(VAS), Oswestry Disability Index(ODI), radiological evidence of intervertebral height and range of motion(ROM) of the treated segment at pre- and post-operation. Operation duration and blood loss was recorded. The clinical outcomes and complications were evaluated afterwards. All patients received a 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria was Single-segmental LDH with low back pain and radicular pain.

Exclusion Criteria:

Exclusion criterias were lumbar stenosis(LSS), lumbar spondylolysis and degenerative spondylolisthesis, spinal deformity, lumbar surgery history, obviously osteoporosis, vertebral fracture, cauda equina syndrome, ankylosing spondylitis, tuberculosis, infection, tumor, obesity.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 2 year
  visual analog scale(0-10 scores) is for pain, 0 represent no pain, 10 score represent the severe pain.
Oswestry Disability Index | 2 year
  Oswestry Disability Index is for movement function, Questionnaire examines perceived level of disability in everyday activities of daily living. The ODI score (index) is calculated as: For example: If all 10 sections are completed, the score is calculated as follows: if 16 (total scored) out of 50 (total possible score) x 100 = 32%; If one section is missed (or not applicable), the score is calculated: If 16 (total scored) / 45 (total possible score) x 100 = 35.5%.
Intervertebral height | 2 year
  Intervertebral height in X-ray is for recontruction of the intervertebral space.
Range of motion(ROM) | 2 year
  ROM was measured by the flexion-extension radiographs of both endplates of the treated segment.